CLINICAL TRIAL: NCT04544878
Title: Clinical and Biological Characteristics of Critically Ill Patients With COVID-19 Admitted to Pediatric Intensive Care Unit
Brief Title: Pediatric Intensive Care and COVID-19
Acronym: CLOVIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Pierre Tissieres, Professor, Bicetre Hospital
Other Study IDs: PS-PICRN--20001
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Covid19; Pediatric ALL; Infection; Critical Illness; SARS-CoV Infection
Keywords: Children; monitoring; immunodepression; HLA-DR; myeloid derived suppressor cell; neutrophil; phenotype
MeSH Terms: conditions — COVID-19; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Infections; Critical Illness; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric patients: All term children from birth to 18 years of age admitted in the PICU
- Adult patients: All patients >18 years of age

SUMMARY:
In this prospective longitudinal cohort the investigators reported the clinical, and biological characteristics of all critically ill patients admitted in the pediatric intensive care unit (PICU) of Bicêtre Hospital during the 2019 coronavirus disease (COVID-19) pandemics. Patients were older than 37 weeks of gestational age. No upper limit was set as the unit was transiently converted into a pediatric "adult COVID-19" intensive care unit.

DETAILED DESCRIPTION:
All patients will be monitored during their PICU stay.

Clinical characteristics include: age, gender, co-morbidities, organ support therapies (mechanical ventilation, renal replacement therapy, extracorporeal membrane oxygenation, vasopressors), organ complications (pulmonary embolism, acute respiratory distress syndrome, renal failure, heart failure) and function, infective complications (ventilator associated pneumonia, central line associated bloodstream infection, pulmonary access, sepsis, septic shock), microbiologic and viral identification, 7-day and 28-day mortality.

Biological characteristics include:

* Admission workup: qualitative and quantitative Ig, ferritin, creatinine kinase, complement study (C3,C4,CH50),
* Daily workup: blood cells count, arterial blood gas analysis, lactate, electrolytes, albumin, blood urea nitrogen, creatinine, hemostasis (fibrinogen, factor V, II+VII, factor X, prothrombin time, antiXa activity, activated cephalin time, D-dimer), C-reactive protein, procalcitonin.
* Twice weekly workup: circulating cells phenotyping (T cell and subclass including Treg, B cell, Natural Killer cell, myeloid derived suppressor cell, neutrophils), interleukin 6.
* Bone marrow analysis when indicated by attending staff.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected or confirmed of severe acute respiratory syndrome Coronavirus 2 infection
* No opposition from patients or legal representatives after study information
* Patients admitted to the pediatric intensive care unit of Bicêtre Hospital, Assistance Publique Hôpitaux de Paris - Paris Saclay University
* Between March 15, 2020 to June 31, 2021

Exclusion Criteria:

* Patient or legal representative refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Most patients admitted in the PICU of Bicêtre Hospital are children <18 years old. Adults critically ill patients with COVID-19 were admitted in case of patients overflow in adult Intensive Care Unit.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-26 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of patient with secondary infection | 2 weeks
  Secondary infection will include healthcare associated infections as well as sepsis, and septic shock

SECONDARY OUTCOMES:
Number of patients dying | 7-day, 28-day and 60-day
  mortality
Description of clinical phenotypes | through study completion, an average of 4 weeks
  Description of the variable clinical phenotypes of COVID-19 in adults and children. This include COVID-19 respiratory failure, acute myocarditis and multi system inflammatory syndrome in children (MIS-C)
Description of immunological phenotypes | through study completion, an average of 4 weeks
  Measure circulating cell phenotypes (relative percentage and monocyte classII histocompatibility complex

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Tissieres, MD, DSc, Principal Investigator — Bicêtre Hospital
Locations (1):
- Pediatric Intensive Care and Neonatal Medicine, Bicêtre Hospital, AP-HP PAris Saclay University, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: Undecided